CLINICAL TRIAL: NCT05675371
Title: A Prospective, Multi-Center, Longitudinal Study of Dynamic Quantification of Social-Visual Engagement (DQSVE) For Treatment Monitoring In Children With Autism Spectrum Disorder (ASD).
Brief Title: Treatment Monitoring in Autism Spectrum Disorder (ASD) in Children
Acronym: MEASURE-ASD1
Status: Completed | Type: Observational
Sponsor: EarliTec Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-1005 (Module 1)
Record Dates: First submitted 2022-12-21; First posted 2023-01-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder; Autism; Developmental Delay; Autism, Early Infantile; Autism, Infantile
Keywords: ASD; autism; autism spectrum disorder; developmental delay; autism in children; autism spectrum disorder in children; autism spectrum disorder in toddlers; autism in toddlers; EarliPoint System: Evaluation for Autism Spectrum Disorder; EarliPoint; DQSVE
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Learning Disabilities | interventions — Applied Behavior Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (4):
- 1a - Typically developing (ages 16-30 months): Typically developing toddlers ages 16 - 30 months (chronological age).
  Interventions: Behavioral: Assessment by Expert Clinician During Behavioral Intervention (ABA or similar); Device: Assessment by the EarliPoint Assessment For Autism Spectrum Disorder
- 1a - ASD/DD (ages 16-30 months): Toddlers ages 16-30 months with autism spectrum disorder and/or related developmental delay who are undergoing applied behavioral analysis (ABA) or related therapies.
  Interventions: Behavioral: Assessment by Expert Clinician During Behavioral Intervention (ABA or similar); Device: Assessment by the EarliPoint Assessment For Autism Spectrum Disorder
- 1b - Typically developing (ages 31-84 months): Typically developing children ages 31-84 months (chronological age).
  Interventions: Behavioral: Assessment by Expert Clinician During Behavioral Intervention (ABA or similar); Device: Assessment by the EarliPoint Assessment For Autism Spectrum Disorder
- 1b - ASD/DD (ages 31-84 months): Children ages 31-84 months with autism spectrum disorder and/or related developmental delay who are undergoing applied behavioral analysis (ABA) or related therapies.
  Interventions: Behavioral: Assessment by Expert Clinician During Behavioral Intervention (ABA or similar); Device: Assessment by the EarliPoint Assessment For Autism Spectrum Disorder

INTERVENTIONS:
Behavioral: Assessment by Expert Clinician During Behavioral Intervention (ABA or similar) — Assessment (e.g., responder vs. non-responder status) utilizing gold-standard clinical reference assessments performed by expert clinicians as the subject undergoes Applied Behavioral Analysis (ABA) or similar intervention for autism spectrum disorder and related developmental delays
  Other Names: Applied Behavior Analysis
Device: Assessment by the EarliPoint Assessment For Autism Spectrum Disorder — Assessment by The EarliPoint™ Evaluation for Autism Spectrum Disorder (ASD), a medical device which employs Dynamic Quantification of Social-Visual Engagement (DQSVE) to aid clinicians in the diagnosis, assessment, and treatment monitoring of ASD related developmental delays, is a diagnostic tool which measures an individual's visual preferential attention to social information in the environment relative to normative age-specific benchmarks.
  Other Names: EarliPoint System: Assessment for Autism Spectrum Disorder

SUMMARY:
The goal of this clinical study is to learn about the utility and performance of the EarliPoint(™) System: Evaluation for Autism Spectrum Disorder to monitor changes in a child's verbal ability, non-verbal learning, and social disability over time in children ages 15-84 months with autism spectrum disorder or related developmental delays (DD) and in those who are typically developing.

The main questions it aims to answer are:

* To estimate the change in each of the EarliPoint index scores in typically developing children ages 15-84 months from baseline through 180 days as a function of the child's age.
* To estimate the change in the EarliPoint verbal and non-verbal index scores in ASD/DD children ages 15-84 months from baseline through 180 days as a function of the child's age in: a) those who showed clinical improvement, and b) those who did not show clinical improvement.
* To estimate the relationship of the EarliPoint verbal and non-verbal index scores to clinical reference assessments in ASD/DD children as a function of their age from baseline through 180 days.
* To estimate the degree of change, if change occurs, month-to-month in the EarliPoint Social Disability Index score from baseline through 180 days.
* To estimate the incidence of behavioral events (e.g., tantrums, etc.) which limit the subject from completing an eye-tracking session.
* To estimate the incidence of adverse device effects associated with the use of the study device.

DETAILED DESCRIPTION:
This study seeks to evaluate the utility and performance of the EarliPoint(™) System: Evaluation for Autism Spectrum Disorder in monitoring changes in a child's verbal ability, non-verbal learning, and social disability over time in children ages 15-84 months with autism spectrum disorder and in those who are typically developing.

The main questions it aims to answer are:

* To estimate the change in each of the EarliPoint index scores in typically developing children ages 15-84 months from baseline through 180 days as a function of the child's age.
* To estimate the change in the EarliPoint verbal and non-verbal index scores in ASD/DD children ages 15-84 months from baseline through 180 days as a function of the child's age in: a) those who showed clinical improvement, and b) those who did not show clinical improvement.
* To estimate the relationship of the EarliPoint verbal and non-verbal index scores to clinical reference assessments in ASD/DD children as a function of their age from baseline through 180 days.
* To estimate the degree of change, if change occurs, month-to-month in the EarliPoint Social Disability Index score from baseline through 180 days.
* To estimate the incidence of behavioral events (e.g., tantrums, etc.) which limit the subject from completing an eye-tracking session.
* To estimate the incidence of adverse device effects associated with the use of the study device.

ELIGIBILITY:
Inclusion Criteria (cohort 1a):

Subjects must meet all the following inclusion criteria to participate in Cohort 1a.

1. Male or female individuals between the ages of 15-30 months (chronological age) at the time of consent who have autism spectrum disorder and/or related developmental delays or those who are typically developing.
2. Normal or corrected-to-normal vision with visual acuity and oculomotor function sufficient to watch short videos.
3. Hearing adequate to hear information presented in age-appropriate videos of social interactions.
4. For individuals who have autism spectrum disorder and/or related developmental delays, the subject must be established in treatment (e.g., a treatment plan has been developed and child is undergoing treatment or will immediately begin treatment) and intends to remain in treatment continuously throughout the duration of the study. Additionally, individuals must provide a diagnostic report documenting a positive diagnosis of ASD/DD available for review. If a report is not available, subjects must undergo diagnostic evaluation prior to enrolling into the study.
5. For individuals who are typically developing, the parent, referring clinician and/or daycare center have indicated that the child is not suspected of, nor has he/she exhibited signs of, developmental delays. NOTE: If, at screening, the investigator suspects the typically developing (TD) subject of having a developmental delay (based on feedback from referring clinician and/or daycare center along with expert clinician opinion), the subject shall be screen failed. He/she should be referred for diagnosis and then may be re-screened for the study.
6. Subject and parent (or legally authorized representative) are able and agree to attend each required study visit and complete the full battery of psychometric assessments and questionnaires (electronically or in-person where required).
7. Subject's parent (or legally authorized representative) can understand information, instructions, and videos presented in the English language.
8. Subject's parent (or legally authorized representative) can read and understand the Informed Consent Form (ICF).
9. Subject's parent (or legally authorized representative) provides written informed consent allowing the child subject to participate in the study. NOTE: where able, the child subject should also provide assent.

Exclusion criteria (cohort 1a):

Subjects who meet any of the following exclusion criteria are not eligible to participate in Cohort 1a:

1. Severe hearing or visual impairment (e.g., congenital nystagmus, congenital cataracts, previous diagnosis of severe hearing deficits by otoacoustic emissions or auditory brainstem response), which in the opinion of the investigator, would limit the child from completing the EarliPoint eye-tracking procedure or clinical reference assessments.

   Note: Corrective lenses are allowable up to a prescription of +/- 5.0.
2. Subject has an uncontrolled seizure disorder.
3. Subject is unable or unwilling to undergo DQSVE testing for up to 15 minutes per assessment (e.g., child has frequent tantrums and tantrums do not subside within 5 minutes).
4. In the opinion of the investigator, the subject and/or parent (or legally authorized representative) are unable, unwilling, or unlikely to comply with all study required procedures and follow-up assessments or to complete the full battery of psychometric assessments (electronically or in-person where required).
5. Subject is receiving or plans to receive any investigational drug or device for the duration of this study.
6. In the opinion of the Investigator, subject is not a suitable candidate for participation in a research study (NOTE: reason must be specified).
7. Typically developing children who have a 1st degree relative with a diagnosis of autism and/or related developmental delay.

Inclusion criteria (module 1b):

Subjects must meet all the following inclusion criteria to participate in this Cohort 1b.

1. Male or female individuals between the ages of 31-78 months (chronological age) at the time of consent who have autism spectrum disorder and/or related developmental delays or those who are typically developing.

   Note: The EarliPoint system is currently configured to monitor children between the ages of 31-84 months. Therefore, at the time of enrollment, participants must be 78 months to facilitate monitoring through 6 months of follow-up.
2. Normal or corrected-to-normal vision with visual acuity and oculomotor function sufficient to watch short videos.
3. Hearing adequate to hear information presented in age-appropriate videos of social interactions.
4. For individuals who have autism spectrum disorder and/or related developmental delays, the subject must be established in treatment (e.g., a treatment plan has been developed and child is undergoing treatment or will immediately begin treatment) and intends to remain in treatment continuously throughout the duration of the study. Additionally, individuals must provide a diagnostic report documenting a positive diagnosis of ASD/DD available for review. If a report is not available, subjects must undergo diagnostic evaluation prior to enrolling into the study.
5. For individuals who are typically developing, the parent, referring clinician and/or daycare center have indicated that the child is not suspected of, nor has he/she exhibited signs of, developmental delays. NOTE: If, at screening, the investigator suspects the TD subject of having a developmental delay (based on feedback from referring clinician and/or daycare center along with expert clinician opinion), the subject shall be screen failed. He/she should be referred for diagnosis and then may be re-screened for the study.
6. Subject and parent (or legally authorized representative) are able and agree to attend each required study visit and complete the full battery of psychometric assessments and questionnaires (electronically or in-person where required).
7. Subject's parent (or legally authorized representative) can understand information, instructions, and videos presented in the English language.
8. Subject's parent (or legally authorized representative) can read and understand the Informed Consent Form (ICF).
9. Subject's parent (or legally authorized representative) provides written informed consent allowing the child subject to participate in the study. NOTE: where able, the child subject should also provide assent.

Exclusion criteria (module 1b):

Subjects who meet any of the following exclusion criteria are not eligible to participate in Cohort 1b:

1. Severe hearing or visual impairment (e.g., congenital nystagmus, congenital cataracts, previous diagnosis of severe hearing deficits by otoacoustic emissions or auditory brainstem response), which in the opinion of the investigator, would limit the child from completing the EarliPoint eye-tracking procedure or clinical reference assessments.

   Note: Corrective lenses are allowable up to a prescription of +/- 5.0.
2. Subject has an uncontrolled seizure disorder.
3. Subject is unable or unwilling to undergo DQSVE testing for up to 15 minutes per assessment (e.g., child has frequent tantrums and tantrums do not subside within 5 minutes).
4. In the opinion of the investigator, the subject and/or parent (or legally authorized representative) are unable, unwilling, or unlikely to comply with all study required procedures and follow-up assessments or to complete the full battery of psychometric assessments (electronically or in-person where required).
5. Subject is receiving or plans to receive any investigational drug or device for the duration of this study.
6. In the opinion of the Investigator, subject is not a suitable candidate for participation in a research study (NOTE: reason must be specified).
7. Typically developing children who have a 1st degree relative with a diagnosis of autism and/or related developmental delay.

Ages: 15 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 15-84 months (at time of enrollment) who have a diagnosis of autism spectrum disorder/related developmental delay and are actively undergoing applied behavioral analysis or related therapy or those who are typically-developing.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Change in EarliPoint Index Scores in typically developing children | 180 days
  To estimate the change in each of the EarliPoint index scores in typically developing children ages 16-30 months form baseline through 180 days as a function of the child's age.
Change in EarliPoint Index Scores in ASD/DD children | 180 days
  To estimate the change in the EarliPoint verbal and nonverbal index scores in ASD/DD children ages 16-30 months from baseline through 180 days as a function of the child's age in a) those who showed clinical improvement, and b) those who did not show clinical improvement.

SECONDARY OUTCOMES:
Relationship of the EarliPoint index scores to clinical reference assessments | 180 days
  To estimate the relationship of the EarliPoint verbal and nonverbal index scores to the Mullen Scales of Early Learning scores in ASD/DD children as a function of their age from baseline though 180-days.
Incidence of behavioral events which limit completion of an eye-tracking session. | 180 days
  To estimate the incidence of behavioral events (e.g., tantrums, inability to calibrate device to child, etc.) which limit the subject from completing an eye-tracking session.
Incidence of adverse device effects associated with use of the study device | 180 days
  To estimate the incidence of adverse device effects associated with the use of the study device.

CONTACTS AND LOCATIONS:
Overall Officials: John Reviere, Study Director — Vice President, Clinical Affairs
Locations (9):
- United States (9):
  - Southwest Autism Research and Resource Center (SARRC), Phoenix, Arizona
  - Cortica - Glendale, Glendale, California
  - Cortica - Marin, San Rafael, California
  - Cortica - Torrance, Torrance, California
  - Cortica - Weslake Village, Westlake Village, California
  - Emory University/Marcus Autism Center, Atlanta, Georgia
  - Munroe-Meyer Institute / University of Nebraska, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - AJ Drexel Autism Institute, Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones W, Klaiman C, Richardson S, Aoki C, Smith C, Minjarez M, Bernier R, Pedapati E, Bishop S, Ence W, Wainer A, Moriuchi J, Tay SW, Klin A. Eye-Tracking-Based Measurement of Social Visual Engagement Compared With Expert Clinical Diagnosis of Autism. JAMA. 2023 Sep 5;330(9):854-865. doi: 10.1001/jama.2023.13295. PMID 37668621
- [Background] Jones W, Klaiman C, Richardson S, Lambha M, Reid M, Hamner T, Beacham C, Lewis P, Paredes J, Edwards L, Marrus N, Constantino JN, Shultz S, Klin A. Development and Replication of Objective Measurements of Social Visual Engagement to Aid in Early Diagnosis and Assessment of Autism. JAMA Netw Open. 2023 Sep 5;6(9):e2330145. doi: 10.1001/jamanetworkopen.2023.30145. PMID 37669054
- See also: EarliPoint Evaluation for Autism Spectrum Disorder — https://www.earlitecdx.com/solutions/